CLINICAL TRIAL: NCT00889369
Title: Duloxetine for the Treatment of Major Depression in Midlife Women: Effects on Brain Structure and Functioning, Mood, and Quality of Life
Brief Title: Duloxetine for Major Depression in Peri-/Postmenopausal Women
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Eli Lilly and Company (Industry); St. Joseph's Healthcare Hamilton (Other); McMaster University (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WHCC2008-2
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2009-06

CONDITIONS: Major Depressive Disorder
Keywords: depression; duloxetine; menopause; imaging; FMRI; Menopausal staging; vasomotor symptoms
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Use of duloxetine, flexible dose (60-120mg/day) for 8 weeks, following a 2-week placebo lead-in phase
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Duloxetine, flexible dose, 60-120mg/per day for 8 weeks, following a 2-week placebo lead-in phase to determine study eligibility
  Other Names: Cymbalta (duloxetine)

SUMMARY:
The main objective of this study is to characterize a range of brain activation symptoms associated with major depression in peri- and post-menopausal women. Also, assessing brain activation before and after the treatment might help to uncover some mechanisms associated with the pathophysiology of depression and menopause.

DETAILED DESCRIPTION:
Women approaching menopause and during the post-menopausal years appear to be at greater risk for developing major depressive episodes. Moreover, this period in life has been associated with significant functional impairment due to the presence/severity of vasomotor symptoms (hot flashes, night sweats), cognitive complaints, and poorer quality of life. In light of recent controversies involving the use of hormone therapies, most physicians and patients are seeking nonhormonal strategies to alleviate menopause-related physical and emotional complaints. Duloxetine has been shown to improve major depressive disorder (MDD) and menopause-related symptoms. To date, the effects of this agent on brain structure and functioning in midlife women with MDD have not been explored. The present study aims to investigate the effects of duloxetine on brain structure and functioning when used for the treatment of a major depressive episode in menopausal women using anatomical magnetic resonance imaging (MRI) and functional MRI (fMRI). In addition, the investigators will examine whether the impact of treatment with duloxetine on vasomotor symptoms, cognition, and quality of life modulate the putative changes in brain structure and functioning.

ELIGIBILITY:
Inclusion Criteria:

* peri-/postmenopausal women, aged 40-60 year
* moderate to severe major depressive episode

Exclusion Criteria:

* DSM-IV Axis I diagnosis other than MDD
* contraindications to magnetic resonance imaging
* treatment-resistent
* previous failed treatment with duloxetine
* history of substance abuse or dependence in past year
* serious suicidal risk
* use of other psychotropic medications
* electroconvulsive therapy or transmagnetic stimulation in past year
* history of allergic reactions to duloxetine
* significant laboratory abnormalities at baseline
* severe hepatic impairment
* end stage renal disease and undergoing dialysis
* uncontrolled narrow-angle glaucoma
* uncontrolled or untreated hyper-/hypothyroidism, or abnormal thyroid stimulating hormone concentration

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-02 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
The effects of response to treatment with duloxetine on brain structure and activation in subjects (peri- and postmenopausal women with MDD). | 10 weeks

SECONDARY OUTCOMES:
Changes in brain activation in remitters versus non-remitters after treatment with duloxetine (remission of depression defined MADRS total score <10 at study end). | 10 weeks
Correlations between changes in brain activation and changes from baseline to study end and menopausal symptoms, depressive symptoms, cognition, quality of life, and clinical global impression (improvement and severity). | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Claudio N Soares, MD, PhD, Principal Investigator — St. Joseph's Healthcare; McMaster University
Locations (1):
- Women's Health Concerns Clinic, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Frey BN, Hall GB, Attard S, Yucel K, Skelin I, Steiner M, Soares CN. Shift in the brain network of emotional regulation in midlife women: is the menopausal transition the turning point? Menopause. 2010 Jul;17(4):840-5. doi: 10.1097/gme.0b013e3181df840f. PMID 20616670